CLINICAL TRIAL: NCT00944008
Title: PROCEDYTE: An Open, Prospective, Multicentre Clinical Trial With Historic Control to Determine Efficacy and Safety of Depocyte® Administration (Liposomal Cytarabine) as Prophylaxis of Neuromeningeal Infiltration of Patients Between 16 and 30 Years Old With Standard Risk Acute Lymphoblastic Leukemia (ALL
Brief Title: PROCEDYTE: Depocyte® Administration (Liposomal Cytarabine) as Prophylaxis of Neuromeningeal Infiltration in Acute Lymphoblastic Leukemia
Acronym: 2009-009422-92
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRODECYTE
Record Dates: First submitted 2009-06-08; First posted 2009-07-22 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia (ALL); Depocyte®; Neuromeningeal relapse; Between 16 and 30 years old; Standard risk
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Depocyte (Experimental)
  Interventions: Drug: DepoCyte

INTERVENTIONS:
Drug: DepoCyte

SUMMARY:
The primary objective is:

* To determine the efficacy and safety of DepoCyte®, as the only intrathecal (IT) prophylaxis of neuromeningeal relapse for patients between 16 and 30 years old diagnosed with acute lymphoblastic leukemia of standard risk treated with the PETHEMA LAL-RI-08 Protocol Chemotherapy schedule.

The secondary objectives are:

* To evaluate the tolerability of IT DepoCyte® as CNS prophylaxis of CNS via IT for patients between 16 and 30 years old with ALL of standard risk.
* To compare the frequency of relapse in CNS for patients between 16 and 30 years old with standard risk ALL treated with the PETHEMA LAL-RI-08 Protocol Chemotherapy schedule and receiving DepoCyte® as the only IT CNS prophylaxis, with that observed in an historic group of patients of identical risk that were treated with the PETHEMA LAL-RI/96 protocol (same systemic chemotherapy and double administration of triple intrathecal chemotherapy)
* To evaluate the frequency of systemic relapses of standard risk ALL patients between 16 and 30 years old treated with the PETHEMA LAL-RI-08 Protocol and who receive DepoCyte® as the only IT prophylaxis of CNS involvement and to compare with those observed in the identical risk patients treated with PETHEMA LAL-RI/96 protocol (same systemic chemotherapy and double administration of triple IT chemotherapy)

DETAILED DESCRIPTION:
A total of 85 patients between 16 and 30 years old with ALL of standard risk will be included in the study. The aim of this study is to determine the efficacy and safety of the administration of DepoCyte® as the only IT prophylaxis of the neuromeningeal relapse in patients between 16 and 30 years old diagnosed with ALL of standard risk.

The study is divided in:

Screening: 2 weeks before treatment Treatment: 2 years of systemic treatment according to PETHEMA LAL-RI-08 Protocol (Induction, Consolidation 1 and 2, Maintenance-1 with reinductions and maintenance 2 with no reinductions). Patients will receive DepoCyte® in Induction, Consolidation 1 and 2 and Maintenance 1 (first year). Patients will not receive DepoCyte® in Maintenance-2 (second year).

Follow-up: Patients in the study will be followed up for one year

ELIGIBILITY:
Inclusion Criteria:

* According to the investigator opinion, patient must able to carry out with all the clinical trial requirements
* Patient or Legal Representative must volunteer sign the inform consent before any study specific test, that is not part of the common patient attention, is performed.
* Age 16 to 30
* Patient diagnosed with standard risk ALL no previously treated. Standard risk ALL is defined by the following criteria:
* Leukocyte count < 25x109/L
* Absence of poor prognosis cytogenetic abnormalities:

  t(9;22) or demonstration of BCR-ABL rearrangements. 11q23 alterations or demonstration of ALL1-AF4 rearrangements.
* Childbearing women must have a negative pregnancy test and must accept to use an effective contraception method.

Exclusion Criteria:

* CNS involvement at diagnosis, defined as presence of blasts in a centrifugated sample of craneospinal fluid with a cellular count of more than 5 cels/L, in the absence of traumatic puncture (more than 10 red blood cels/ml), or as neurological symptoms that suggest of neuromeningeal involvement and imaging tests compatible, in the absence of blasts in craneospinal fluid.
* B mature cell phenotype (sIg+) or with the Burkitt ALL cytogenetic abnormalities (t[8;14], t[2;8], t[8;22])
* ALL with t(9;22) or BCR-ABL rearrangements.
* Acute biphenotypic and bilineal leukemias
* Acute undifferentiated leukemia
* History of coronary or valvular disease or hypertensive cardiopathy
* Chronic hepatopathy
* Chronic respiratory insufficiency
* Chronic renal insufficiency not due to ALL
* Serious neurological disorders not due to ALL
* Abnormal ECOG (WHO scale grade 3 and 4) not done by ALL
* Pregnant or currently breast feeding women
* Patients participating in other clinical trial or receiving any other investigational agent within 30 days previous to the study inclusion

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of DepoCyte®, as the only intrathecal (IT) prophylaxis of neuromeningeal relapse | 1 year

SECONDARY OUTCOMES:
Tolerability of IT DepoCyte | 2 months
Compare the frequency of relapse in CNS with an historic group of patients of identical risk that were treated with the PETHEMA LAL-RI/96 protocol | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sancho Jose Manuel, Dr, Study Chair — Germans Trias i Pujol Hospital
Locations (17):
- Spain (17):
  - Hoapital General, Alicante
  - Hospital Clínic, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital vall d'Hebrón, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico, Madrid
  - Hospital La Paz., Madrid
  - Hospital Carlos Haya., Málaga
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer., Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Son Dureta., Palma de Mallorca
  - Hospital Clínico Universitario, Salamanca
  - Hospital Universitario Virgen del Rocío., Seville
  - Hospital clínico Universitario, Valencia

REFERENCES:
- See also: Spanish Asotiation of Hematology — http://aehh.org